CLINICAL TRIAL: NCT04081077
Title: Pharmacokinetics and Pharmacodynamics Sub-study for TB-PRACTECAL Clinical Trial ( PRACTECAL-PKPD)
Brief Title: PRACTECAL-PKPD Sub Study
Acronym: PRACTECAL-PKPD
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medecins Sans Frontieres, Netherlands (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Global Alliance for TB Drug Development (Other); University College, London (Other); Drugs for Neglected Diseases (Other); Swiss Tropical & Public Health Institute (Other); eResearch Technology, Inc. (Industry); Ministry of Health, Republic of Uzbekistan (Other Government); World Health Organization (Other); Ministry of Public Health, Republic of Belarus (Other Government); THINK TB & HIV Investigative Network (Network); University of Liverpool (Other); Wits Health Consortium (Pty) Ltd (Other); Hackensack Meridian Health (Other); University of California, San Francisco (Other); Minsk Republican Research and Practical Centre for Pulmonology and Tuberculosis (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRACTECAL-PKPD
Record Dates: First submitted 2019-08-29; First posted 2019-09-09 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Multi-drug Resistant Tuberculosis; Extensively Drug-Resistant Tuberculosis; Pulmonary Tuberculosis
Keywords: Pharmacokinetics; Pharmcogenomics; Pharmacodynamics; Bedaquiline; Pretomanid; Linezolid; Clofazimine; Moxifloxacin
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Extensively Drug-Resistant Tuberculosis; Tuberculosis, Pulmonary | interventions — bedaquiline; pretomanid; Moxifloxacin; Linezolid; Clofazimine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regimen 1: Bedaquiline, Pretomanid, Linezolid, Moxifloxacin (Experimental): Bedaquiline: 400 mg once daily for 2 weeks followed by 200 mg 3 times per week for 22 weeks Pretomanid: 200mg once daily for 24 weeks Moxifloxacin: 400 mg once daily for 24 weeks Linezolid: 600mg daily for 16 weeks then 300mg daily (or 600mg x3/wk) for the remaining 8 weeks or earlier when moderately tolerated
  Interventions: Drug: Bedaquiline; Drug: Pretomanid; Drug: Moxifloxacin; Drug: Linezolid
- Regimen 2:Bedaquiline, Pretomanid, Linezolid, Clofazimine (Experimental): Bedaquiline: 400 mg once daily for 2 weeks followed by 200 mg 3 times per week for 22 weeks Pretomanid: 200mg once daily for 24 weeks Linezolid: 600mg daily for 16 weeks then 300mg daily (or 600mg x3/wk) for the remaining 8 weeks or earlier when moderately tolerated Clofazimine: 50 mg (less than 33 kg), 100 mg (more than 33 kg) for 24 weeks
  Interventions: Drug: Bedaquiline; Drug: Pretomanid; Drug: Linezolid; Drug: Clofazimine
- Regimen 3: Bedaquiline, Pretomanid, Linezolid (Experimental): Bedaquiline: 400 mg once daily for 2 weeks followed by 200 mg 3 times per week for 22 weeks Pretomanid: 200mg once daily for 24 weeks Linezolid: 600mg daily for 16 weeks then 300mg daily (or 600mg x3/wk) for the remaining 8 weeks or earlier when moderately tolerated)
  Interventions: Drug: Bedaquiline; Drug: Pretomanid; Drug: Linezolid

INTERVENTIONS:
Drug: Bedaquiline — Bedaquiline is a diarylquinoline class antimicrobial which blocks the proton pump for ATP synthase of mycobacteria. This in turn blocks the ATP production required for cellular energy production and leading to cell death.
  Other Names: Sirturo; R207910; TMC207
Drug: Pretomanid — Pretomanid is an nitroimidazole class antimicrobial which interferes with cell wall biosynthesis in mycobacteria. It may have other mechanisms of action as well in non-replicating mycobacteria.
  Other Names: PA-824
Drug: Moxifloxacin — Moxifloxacin is an 8-methoxyquinolone class antimicrobial that is a potent inhibitor of DNA gyrase and topoisomerase IV in bacteria
  Other Names: Avelox, BAY 12-8039
  Arms: Regimen 1: Bedaquiline, Pretomanid, Linezolid, Moxifloxacin
Drug: Linezolid — Linezolid, an oxazolidinone class antimicrobial which works by inhibiting ribosomal protein synthesis. It is approved for Gram-positive bacterial infections, and is increasingly being used for drug resistant TB disease.
  Other Names: Zyvox
Drug: Clofazimine — Clofazimine (Cfz) is a lipophilic riminophenazine licensed for treatment of leprosy. Its mechanism(s) of action remains unclear, but existing evidence suggests production of reactive oxygen species within Mycobacterium tuberculosis is one mechanism.
  Other Names: Lamprene
  Arms: Regimen 2:Bedaquiline, Pretomanid, Linezolid, Clofazimine

SUMMARY:
PRACTECAL-PKPD is an exploratory pharmacokinetic and pharmacodynamic sub-study investigating the relationship between the patients' exposure to anti- tuberculosis (TB) drugs in the TB-PRACTECAL trial investigational regimens and their respective treatment outcomes.

DETAILED DESCRIPTION:
PRACTECAL-PKPD is a sub-study of the main TB-PRACTECAL phase II-III trial for the treatment of biologically confirmed pulmonary multi drug or extensively drug-resistant TB (M/XDR-TB). TB-PRACTECAL is a multicentre, open label, phase 2-3 randomised controlled trial evaluating 6 months, exclusively oral regimens containing bedaquiline (B), pretomanid (Pa), linezolid (Lzd) +/- moxifloxacin (Mfx) or clofazimine (Cfz) for the treatment of microbiologically confirmed pulmonary M/XDR-TB.

Primary objective Measure the plasma concentrations of pretomanid, linezolid, bedaquiline, clofazimine and moxifloxacin in a sub-set of patients in the TB-PRACTECAL trial and using population pharmacokinetic (PK) models, estimate the population exposure metrics (minimum plasma concentration (Cmin), mean plasma concentration (Cmean), maximum plasma concentration (Cmax), plasma concentration versus time curve (AUC)) for the individual drugs in the TB-PRACTECAL trial.

Secondary objectives Develop a population pharmacodynamic model to explore the relationship between drug exposure, baseline minimum inhibitory concentrations and both mycobacteriological and clinical treatment success Develop a population pharmacodynamics model and identify PK parameters that are associated with treatment emergent toxicity Explore covariates specific to the regimens and study population Use results of above objectives to develop a hypothesis on the optimal dosing of linezolid and clofazimine Explore the pharmacogenomic factors associated with efficacy and toxicity of the investigational drugs Analyse adherence/exposure to the investigational regimen(s) by analysing anti-TB drug levels in small hair samples Assess the potential of using hair drug levels to develop safety and efficacy pharmacodynamic models Conduct clinical validation of a dried blood quantification method using volumetric absorptive microsampling.

Procedures:

4 ml (vacutainer tube, lithium heparin) of blood will be collected from the hand, forearm or antecubital vein at each sampling occasion and moment for the PK. The sampling occasions are on Day 1, Weeks 8, 12, 16, 20, 24, 32 and 72. On Day 1, blood will be collected just before drugs intake, then 2 and 23 hours after drugs intake. On week 8, blood will be collected just before drugs intake, then 6.5 and 23 hours post dose. At weeks 12, 16, 20 and 24 the blood will be collected within 30 minutes before taking the dose. Samples from week 32 and 72 will be collected whenever feasible after the patients have completed their treatment so blood collection is not relative to drug intake on that occasion. These have been included to capture the elimination phases of the drugs which have long terminal half-lives.

A subgroup of patients will also participate to the clinical validation study of a dried blood quantification method using volumetric absorptive microsampling. 2ml of blood and a drop of blood from the finger tips will be collected at the following sampling occasions: day 1, week 8, 12 and 16.

In the small hair study, a small thatch of hair will be cut as close as possible to the scalp from the occiput at weeks 8, 16, 24, 32 and 72.

ELIGIBILITY:
Main study inclusion criteria*:

Patients eligible for inclusion in the trial must fulfil all of the following criteria:

* Male or female subjects aged 15 years of age or above, regardless of HIV status;
* Microbiological test (molecular or phenotypic) confirming presence of M. tuberculosis;
* Resistant to at least rifampicin by either molecular or phenotypic drug susceptibility test;
* Completed informed consent form (ICF);

Main study exclusion criteria:

* Known allergies, hypersensitivity, or intolerance to any of the study drugs;
* Pregnant or breast-feeding; or unwilling to use appropriate contraceptive measures
* Liver enzymes >3 times the upper limit of normal;
* Any condition (social or medical) which, in the opinion of the investigator, would make study participation unsafe;
* Taking any medications contraindicated with the medicines in the trial; QTcF > 450ms;
* One or more risk factors for QT prolongation (excluding age and gender) or other uncorrected risk factors for TdP;
* History of cardiac disease, syncopal episodes, symptomatic or asymptomatic arrhythmias (with the exception of sinus arrhythmia);
* Any baseline biochemical laboratory value consistent with Grade 4 toxicity.
* Moribund
* Known resistance to bedaquiline, pretomanid, delamanid or linezolid.
* Prior use of bedaquiline and/or pretomanid and/or linezolid and/or delamanid for one or more months.
* Patients not eligible to start a new course of MDR-TB/XDR-TB treatment according to local protocol, including but not limited to:

  * currently on MDR-TB treatment for more than 2 weeks (and not failing)
  * unstable address
  * loss to follow-up in previous treatment with no change in circumstance and motivation.
* Tuberculous meningoencephalitis, brain abscesses, osteomyelitis or arthritis.

  *PKPD inclusion/exclusion:
* Adult patients (aged 18 years or above) recruited into the investigational arms of the TB-PRACTECAL trial in the approved sites.
* Willing to sign the sub-study informed consent form after agreeing to the additional blood draws.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-08-06 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic: Cmax | 72 weeks
  Plasma concentrations, their timing in relation to dose intake and start of treatment will be used in a population PK model to estimate Peak Plasma Concentration (Cmax)
Pharmacokinetic: AUC | 72 weeks
  Plasma concentrations, their timing in relation to dose intake and start of treatment will be used in a population PK model to estimate the area under the plasma concentration versus time curve (AUC)
Pharmacokinetic: T1/2 | 72 weeks
  Plasma concentrations, their timing in relation to dose intake and start of treatment will be used in a population PK model to estimate the elimnation half life (T1/2)
Pharmacokinetic: Tmax | 72 weeks
  Plasma concentrations, their timing in relation to dose intake and start of treatment will be used in a population PK model to estimate the time present at maximum plamsa concentration (Tmax)
Pharmacodynamics: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 72 weeks
  Number of patients with serious adverse events (SAE), adverse events of special interest (AESI) and other AEs with their respective severity grading.
Pharmacodynamics: Culture Conversion 24 weeks post treatment [Efficacy] | 24 weeks
  Percentage of patients with culture conversion in liquid media at 24 weeks post randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Bern Nyang'wa, MB BS, MPH, Principal Investigator — Medecins Sans Frontieres, Netherlands
Locations (5):
- Republican Scientific and Practical Centre for Pulmonology and Tuberculosis hospital, Minsk, Belarus
- South Africa (4):
  - Helen Jospeh Hospital, Johannesburg, Gauteng
  - THINK Clinical Trial Unit, Hillcrest, Durban, KwaZulu-Natal
  - King DinuZulu Hospital, Durban, KwaZulu-Natal
  - Doris Goodwin Hospital, Pietermaritzburg, KwaZulu-Natal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nyang'wa BT, Kloprogge F, Moore DAJ, Bustinduy A, Motta I, Berry C, Davies GR. Population pharmacokinetics and pharmacodynamics of investigational regimens' drugs in the TB-PRACTECAL clinical trial (the PRACTECAL-PKPD study): a prospective nested study protocol in a randomised controlled trial. BMJ Open. 2021 Sep 6;11(9):e047185. doi: 10.1136/bmjopen-2020-047185. PMID 34489274